CLINICAL TRIAL: NCT02482935
Title: The Effect of Food on the Pharmacokinetics of the Proposed Commercial Formulation of Abemaciclib in Healthy Subjects
Brief Title: A Study of Abemaciclib (LY2835219) in Healthy Participants With and Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15536; I3Y-MC-JPBU (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abemaciclib High Fat Meal (Experimental): Abemaciclib capsules administered once orally in the fed state.
  Interventions: Drug: Abemaciclib
- Abemaciclib Fasted (Experimental): Abemaciclib capsules administered once orally in the fasted state.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The purpose of this study is to evaluate the amount of abemaciclib that reaches the blood stream and how long the body takes to get rid of it when given with and without food. In addition, the safety and tolerability of the study drug will be evaluated. Information about any side effects that may occur will also be collected. The study will last about 43 days for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy sterile males or surgically sterile or postmenopausal females
* Have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m^2), inclusive

Exclusion Criteria:

* Participated in a clinical trial involving investigational product within 30 days
* Have known allergies to abemaciclib, related compounds or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure
* Show evidence of human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to stop alcohol consumption 48 hours prior to each admission until collection of the last PK sample in each period
* Are unwilling to refrain from consuming xanthine-containing food and drink from 48 hours prior to admission until collection of the last pharmacokinetic (PK) sample in each period
* Are currently or have been smokers or users of tobacco or nicotine replacement products within the 6 months prior to admission or have a positive urine cotinine test
* Are unwilling to comply with the dietary requirements/restrictions during the study: Consume only the meals provided during the inpatient stays and refrain from eating any food or drinking any beverages containing grapefruit, grapefruit juice, grapefruit-containing products, Seville oranges, star fruit or star fruit juice, pomelo, or commercial apple juice or orange juice for at least 2 weeks prior to the first dose until the final PK sample is collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this two-period crossover study, abemaciclib was administered once (fasting or fed) in each period. There were at least 16 days between doses and follow-up was completed 15 to 18 days after the last dose in Period 2.
Groups:
- Abemaciclib Fasted/Fed: 200 milligrams (mg) abemaciclib administered orally, once in a fasted state, then once in a fed state.
- Abemaciclib Fed/Fasted: 200 mg abemaciclib administered orally, once in a fed state, then once in a fasted state.
Period: Period 1
Arm/Group | Abemaciclib Fasted/Fed | Abemaciclib Fed/Fasted
Started | 15 | 15
Received Abemaciclib | 15 | 15
Washout | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Abemaciclib Fasted/Fed | Abemaciclib Fed/Fasted
Started | 14 | 15
Received Abemaciclib | 14 | 15
Follow-up | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received abemaciclib.
Groups:
- Abemaciclib: 200 mg abemaciclib administered once orally in each of two study periods.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC [0-inf]) for Both Fed and Fasted Periods for Abemaciclib and Major Metabolites
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 Hours Postdose in Each Period
Population: All participants who received abemaciclib and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms x hours/mililiters (ng·h/mL)
Groups:
- Abemaciclib Fasted: 200 mg abemaciclib administered once, orally, in a fasted state.
- Abemaciclib Fed: 200 mg abemaciclib administered once, orally, in a fed state.
Arm/Group | Abemaciclib Fasted | Abemaciclib Fed
Number analyzed (Participants) | 27 | 29
nanograms x hours/mililiters (ng·h/mL)
  Abemaciclib | 3940 (34) | 4950 (42)
  LSN2839567 | 1630 (27) | 1910 (28)
  LSN3106726 | 3180 (25) | 3410 (28)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) for Both Fed and Fasted Periods for Abemaciclib and Major Metabolites
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 Hours Postdose in Each Period
Population: All participants who received abemaciclib and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Abemaciclib Fasted | Abemaciclib Fed
Number analyzed (Participants) | 28 | 29
ng/mL
  Abemaciclib | 116 (36) | 159 (38)
  LSN2839567 | 33.4 (36) | 41.4 (29)
  LSN3106726 | 55.7 (31) | 61.0 (29)

3. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) for Both Fed and Fasted Periods for Abemaciclib and Major Metabolites
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, and 192 Hours Postdose in Each Period
Population: All participants who received abemaciclib and had evaluable plasma values.
Measure: Median (Full Range); unit: hours
Arm/Group | Abemaciclib Fasted | Abemaciclib Fed
Number analyzed (Participants) | 28 | 29
hours
  Abemaciclib | 8.00 [6.00 to 12.00] | 8.00 [6.00 to 12.00]
  LSN2839567 | 6.00 [3.00 to 12.00] | 6.00 [4.00 to 12.00]
  LSN3106726 | 8.02 [6.00 to 24.02] | 10.00 [6.00 to 24.03]

ADVERSE EVENTS:
Description: All participants who received abemaciclib.
Arm/Group | Abemaciclib Fasted | Abemaciclib Fed
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 4/30 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib Fasted (N=30) | Abemaciclib Fed (N=29)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days